CLINICAL TRIAL: NCT06272591
Title: Comparison of Patient Satisfaction With Home Induction and In-patient Induction.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1192023/CHUSTE
Record Dates: First submitted 2024-01-15; First posted 2024-02-22 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Induced; Birth; Pregnancy
Keywords: Induced labour; Induction of labour; Cervical ripening; Inducing labour at home; Patient's choice of induction method; Experiences induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with induction indication: Any pregnant woman, with a singleton pregnancy, giving birth at Saint-Etienne University Hospital, with an indication for induction of labour from 37SA will be included. The indications may be for a maternal pathology, a maternal wish or a foetal pathology.
  Interventions: Other: Preliminary search in the patient's file; Other: A posteriori research in the patient's file; Other: First questionnaire : choice of induction method reason for choice; Other: Second questionnaire : experience of induction

INTERVENTIONS:
Other: Preliminary search in the patient's file — Details of the information previously sought in the patient's file :
  age profession gender/parity physiological or pathological pregnancy indication for induction of labour gestational age at time of induction
Other: A posteriori research in the patient's file — Data on maternal and foetal morbidity and mortality following childbirth will be collected.
Other: First questionnaire : choice of induction method reason for choice — Given on arrival at the maternity unit to begin induction.
Other: Second questionnaire : experience of induction — Given post-partum in the maternity unit.

SUMMARY:
Induced labour is a medical intervention designed to initiate or accelerate the childbirth process when clinically indicated.

Induced labour concerns 25.8% of pregnant women in France, according to the latest National Perinatal Survey 2021. This rate is rising steadily, since in 2016 induction concerned 22% of pregnancies. There are many medical indications for induction, both maternal and foetal. Induced labour in hospitals is beginning to reach its limits, given the reduction in the number of nursing staff and the reduction in the number of beds available. In some cases, patients are hospitalised for 24 to 72 hours before going into labour. In this context, the place where the birth takes place, whether at home or in hospital, is essential, with a potential impact on patient satisfaction and the experience of induction.

Cervical ripening can be a difficult experience for women, with a feeling of loss of control at this crucial stage. The duration of induction is one of the factors that women would like to see changed when asked about the aftermath of induction. The option of inducing at home might seem to improve women's experience and reduce the length of their stay in hospital.

DETAILED DESCRIPTION:
There are generally two main methods of cervical ripening, mechanical methods (Foley® catheter or Cook® double balloon catheter) and pharmacological methods (Propess® dinoprostone intravaginal tampon, Prostine® intravaginal gel, or Angusta® oral misoprostol).

Balloon induction of labour works by the dilating effect of a balloon inflated at the level of the uterine cervix, which distinguishes it from pharmacological methods acting via uterine contractions.

Balloon induction has been shown to be effective and safe. It therefore seems important to take a closer look at this method of outpatient induction, especially as the risks of uterine hyperkinesia/hypertonia and anomalies in foetal heart rate are very low with this technique.

Several foreign studies have looked at outpatient induction of labour. Meta-analyses have shown a lower caesarean section rate with outpatient induction, faster labour and less administration of oxytocin.

In terms of safety, a systematic review of the literature based on data from 26 studies, published in 2018, showed a low risk of developing adverse effects between insertion and expulsion of the balloon. A meta-analysis conducted in 2020 compared inpatient versus outpatient induction of labour, showing no significant differences between the home and inpatient groups in terms of major neonatal adverse events. In addition, several studies have suggested that allowing patients to participate actively in the decision concerning the induction method can promote better understanding and acceptance of the process, thereby strengthening their commitment to their own health.

The obstetrics and gynecology department of the University hospital recently modified its protocol for the management of induced labour in order to allow a more free and informed choice of technique (information booklet, reflection period) and a return home for low-risk women after balloon insertion.

The aim of this work will be to demonstrate a link between women's choice of induction method and increased compliance with their care.

The aim of this study is to monitor the implementation of this new service protocol.

The aim of the study will be to analyse the experience and satisfaction of women who have undergone induction, comparing their experiences at home and in hospital.

This research is being carried out in a context in which the choice of induction, the methods used and the place of delivery are arousing growing interest in the medical community and among women themselves.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Singleton pregnancy
* Indication for induction of labour ≥ 37SA+0d
* Unfavourable cervix (Bishop<6)
* Living less than 30 minutes' drive from hospital
* Having a relative at her side for a return home

Exclusion Criteria:

* Scarred uterus : previous caesarean section or myomectomy
* Premature rupture of membranes
* Fetal death in utero
* Placenta previa/accreta/percreta
* Severe maternal pathology : decompensated respiratory, cardiac, hepatic, renal, digestive or psychiatric disease, severe pre-eclampsia, severe growth retardation or anamnios
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any pregnant woman with a singleton pregnancy, giving birth at the Saint-Etienne University Hospital, with an indication for induction of labour from 37SA. The indications could be for a maternal pathology, a maternal wish or a foetal pathology.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire on patients' experience of induction in hospital and at home. | Day 2
  To compare patients' experiences of their induction in hospital or at home, using a questionnaire handed out after the birth.
Questionnaire on patients' satisfaction of induction in hospital and at home. | Day 2
  To compare patients' satisfaction of their induction in hospital or at home, using a questionnaire handed out after the birth.

SECONDARY OUTCOMES:
Questionnaire on patients' choice of induction method | Day 0
  To analyse patients' choice of induction method and the reasons for it, using a questionnaire handed out on arrival at the maternity unit.
Questionnaire on reasons for choosing home induction. | Day 0
  Analyse the reasons for choosing home induction based on the answers to the questionnaire given on arrival at the maternity unit.
Maternal morbidity | Day 3
  To compare maternal morbidity between home and hospital induction.
Maternal mortality | Day 3
  To compare maternal mortality between home and hospital induction.
Neonatal morbidity | Day 3
  To compare neonatal morbidity between home and hospital induction.
Neonatal mortality | Day 3
  To compare neonatal mortality between home and hospital induction.

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine BARJAT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No